CLINICAL TRIAL: NCT05491681
Title: Phase I/IIa Study to Assess AllogeneiC Expanded Human Mesenchymal Stem Cell Therapy in Patients Recovering From COVID-19 Acute Respiratory Distress Trial (ACE CARD TRIAL)
Brief Title: AllogeneiC Expanded Human MSC Therapy in Patients Recovering From COVID-19 Acute Respiratory Distress Trial
Acronym: ACE_CARD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: With available funding it was necessary for Sponsor to prioritize other studies. No study participants were consented or enrolled and no study sites were activated.
Sponsor: BioCardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 05539-A
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Dose finding study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): Experimental: Cohort 1 Low dose, 20M cells, 3 patients
  Interventions: Biological: intravenous delivery of allogeneic bone marrow-derived MSCs
- Medium dose (Experimental): Experimental: Cohort 2 Med dose, 100M cells, 3 patients
  Interventions: Biological: intravenous delivery of allogeneic bone marrow-derived MSCs
- High dose (Experimental): Experimental: Cohort 3 High dose, 200M cells, 3 patients
  Interventions: Biological: intravenous delivery of allogeneic bone marrow-derived MSCs

INTERVENTIONS:
Biological: intravenous delivery of allogeneic bone marrow-derived MSCs — MSCs
  Other Names: allogeneic NK1R+MSC

SUMMARY:
Allogeneic culture-expanded bone marrow-derived human mesenchymal stem cells (MSC) are the subject of the current study as they are supported by preclinical and clinical data for potential to provide a safe and effective treatment for patients with acute respiratory distress.

DETAILED DESCRIPTION:
The majority of Covid-19 cases either are asymptomatic or result in only mild disease. However, in a substantial percentage of patients, a respiratory illness requiring hospital care develops, and such infections can progress to critical illness with hypoxemic respiratory failure requiring prolonged ventilatory support (Zhou 2020) , (Chen 2020) , (Cao 2020) , (Ruan 2020) . Among patients with Covid-19 who have been admitted to hospitals in the United Kingdom, the case fatality rate has been approximately 26%, a percentage that has increased to more than 37% among patients who were undergoing invasive mechanical ventilation.(Docherty 2020) Although remdesivir has been shown to shorten the time until recovery in hospitalized patients, (Beigel 2020). Efforts to modulate inflammation-mediated lung injury and thereby reduce progression to respiratory failure and death have shown promising results.

INVESTIGATIONAL PRODUCT The NK1R+ MSC cell therapy are allogeneic bone marrow-derived mesenchymal stem cells that will be delivered intravenously.

Details on cell culture and expansion of the cells are provided in the Chemistry Manufacturing and Controls Section of the IND.

Cells are provided cryopreserved and are thawed, washed, and prepared for IV delivery.

STUDY OBJECTIVES The objective of this clinical trial is to determine the safety and the optimal cell dose of the NK1R+ hMSC in patients recovering from ARDS.

.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years and ≤ 80 at age at consent
2. Patient must have:

   * Have a laboratory-confirmed COVID-19 diagnosis (nucleic acid-based assay (e.g., RTPCR) to establish the diagnosis of SARS-CoV-2 infection), who recovered from moderate to severe COVID-19 associated ARDS, as determined by Berlin Criteria and been weaned off the ventilator support."
   * Meet the criteria for mild and moderate COVID-19 as described in COVID-19: Developing Drugs and Biological Products for Treatment or Prevention Guidance for Industry (Feb 2021).
   * Recovery from moderate to severe ARDS, diagnosed based on Berlin Criteria, within past 7 days.
3. PaO2/FiO2 > 100 to <200 mmHg with PEEP>5cm H2O
4. Patient or legally authorized representative (LAR) provides written informed consent, except as noted in 21 CFR 50.23
5. Understands and agrees to comply with planned study procedures
6. Available for clinical follow-up for duration of the treatment and follow-up period
7. Woman of childbearing potential must have a negative pregnancy test at admission or within 24 hours before starting treatment
8. Agree not to become pregnant during treatment and for 1 months after receiving treatment
9. Use at least 2 reliable forms of effective contraception, including 1 barrier method, during treatment and for 1 month after the treatment period

Exclusion Criteria:

1. Severe chronic respiratory disease with a PaCO2 > 50 mm Hg or the use of home oxygen (chronic obstructive pulmonary disease or pulmonary fibrosis)
2. Be an organ transplant recipient
3. ALT/AST ≥ 5 times the upper limit of normal
4. BMI > 40
5. Stage 4 severe kidney disease or requiring dialysis (i.e. eGFR <30)
6. Anticipated transfer to another hospital that is not a study site within 72 hours
7. Shock or on ECMO
8. Pregnant or nursing
9. On a ventilator at the time of enrollment
10. Have received high dose corticosteroids at doses >20 mg per day (or prednisone equivalent) administered for ≥14 consecutive days in the month prior to study entry.
11. Have been diagnosed with cancer
12. Demonstrated inability to comply with the study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-04 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-01-04 (Actual)

PRIMARY OUTCOMES:
Number of product related adverse events through the duration of the study. | 3 months
  Number of product related adverse events through the duration of the study.

SECONDARY OUTCOMES:
Secondary Endpoint | 12 months
  Number of participants with resolution and/or improvement of ARDS at 7 days, 14 days, 21 days, and 28 days according to the Berlin Criteria.
  * Change in PF ratio from baseline to >200-300, and above >300
  * Absolute change in PF ratio

IPD SHARING:
Plan to Share IPD: No